CLINICAL TRIAL: NCT00580749
Title: Feeding and Pancreatic Rest in Acute Pancreatitis
Brief Title: Study of Nutrition in Acute Pancreatitis
Acronym: SNAP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: not meeting enrollment criteria
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, David Whitcomb, MD, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO 07080011, PRO 07080044; 1 R01 DK 075803-01A1 NIH#
Record Dates: First submitted 2007-12-21; First posted 2007-12-27 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2013-06

CONDITIONS: Pancreatitis
Keywords: Pancreatitis; enteral feeding; distal jejunal feeding; naso gastric feeding; pancreatic rest
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DJ (Active Comparator): Naso disal jejunal(DJ) feedings randomized to 50% of subjects meeting criteria.
  Interventions: Procedure: Naso jejunal feeding tube insertion
- NG (Active Comparator): Placement of naso gastric feeding tube through nare into stomach for enteral feeding.
  Interventions: Procedure: NG feeding tube insertion

INTERVENTIONS:
Procedure: Naso jejunal feeding tube insertion — Placement of feeding tube through nare and into jejunum for administration of enteral feeding.
  Arms: DJ
Procedure: NG feeding tube insertion — Placement of naso gastric feeding tube into stomach for purpose of enteral feedings.
  Arms: NG

SUMMARY:
We will compare the two types of enteral (intestinal) nutrition in regard to patients with severe acute pancreatitis in our institution and also in 8 others in the United States.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over the age of 18yr
2. The typical history of abdominal pain for over 24h with raised (>3-fold) serum pancreatic enzymes on admission
3. Severe pancreatitis, as defined by: the Atlanta classification of severe disease (60), but with important modifications to sharpen the definition of severity, to include one or more of the following:

   1. The presence of organ failure (MOF) resistant to early aggressive IV fluid resuscitation as defined by a Marshall score of ≥2 in any one organ (for calculation, see Appendix (61)), excluding the liver component as the abnormality may be due to gall stones rather than the systemic inflammatory response (17)
   2. Pancreatic necrosis >30% on CT scan or a modified CT severity index (CTSI: see Appendix (62)) of ≥8
   3. APACHE score ≥ 8 (for calculation, see Appendix (63))
   4. Ranson's criteria ≥3 (for calculation, see Appendix (64))

Exclusion Criteria:

1. Inability to absorb enteral nutrients resulting in chronic intestinal failure and need for IV feeding, such as short bowel, malabsorption disorders such as celiac or intestinal proliferative disorders, chronic obstruction and pseudo-obstruction.
2. Time elapse since commencement of acute pancreatitis symptoms >10 days. In order to take advantage of the 'window of opportunity' to prevent the progression of 'transient' MOF to 'permanent' MOF, patients should be started on enteral feeding as soon as possible. However, in practice many patients present initially with mild disease which progresses to severe necrosis at the end of the first week, and these patients need nutritional support for long periods of time. Consequently, this is an important group to include in this investigation. Post hoc analysis will be performed to see whether they behave differently to patients fed earlier in their disease
3. Any form of artificial feeding since commencement of acute pancreatitis symptoms
4. Patients with chronic pancreatitis and pancreatic insufficiency requiring pancreatic enzyme supplements, based on clinical history and specific investigations such as by ERCP, MRP, or CT scanning.
5. Pre-existing chronic renal insufficiency requiring hemodialysis or peritoneal dialysis, as this will make assessment of severity difficult
6. Pre-existing end-stage liver disease with ascites, coagulopathy and encephalopathy, supported by biopsy, and/or radiological imaging and endoscopy (portal hypertension, varices and gastropathy), as this will make assessment of severity difficult
7. Chronic immunodeficiency states such as AIDS defined by CD-4 count < 50, and immunoglobulin deficiencies as it may independently affect feeding tolerance and infection risk
8. Pancreatic cancer proven by biopsy, and any other form of cancer with life-expectancy <6 months.
9. Current somatostatin or corticosteroid therapy as these drugs will impair intestinal, metabolic, and immune function, and therefore affect absorption and infection risk.
10. Contraindication to using the nose for enteral tube insertion
11. Severe traumatic brain injury with ICP>20mmHg despite treatment
12. Previous completion or withdrawal from this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Feeding success as determined by the quantity of nutrition delivered and the number of interruptions due to intolerance and how the two forms of feeding influence disease outcome as measured by duration of ICU and hospital stay. | Approx. one week

SECONDARY OUTCOMES:
Feeding tolerance (nitrogen balance, stool volume, incidence of nausea, incidence of nausea and vomiting) will demonstrate better tolerance for subjects undergoing DJ feeding than those undergoing NG feeding. | Approx. one week

CONTACTS AND LOCATIONS:
Overall Officials: David Whitcomb, MD, Principal Investigator — University of Pittsburgh
Locations (4):
- United States (4):
  - University of Alabama, Birmingham, Alabama
  - University of Florida College of Medicine, Gainesville, Florida
  - Indiana University, Indianapolis, Indiana
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania